CLINICAL TRIAL: NCT05225142
Title: Modified Minimally Invasive Surgical Technique in Human Intrabony Defects With or Without Regenerative Materials 10-year Follow-up of a Randomized Clinical Trial: Tooth Retention, Periodontitis Recurrence and Costs
Brief Title: 10 Year Follow up of RCT Comparing Different Regenerative Regenerative Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The European Research Group on Periodontology (ERGOPerio) (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATRO M-MIST
Record Dates: First submitted 2022-01-25; First posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — emerin

STUDY DESIGN:
Intervention Model Description: Long term follow up of RCT
Who Masked: Investigator, Outcomes Assessor
Masking Description: Allocation concealment of surgeon until completion of common part of surgical intervention. Examiner (clinical and radiographic ) and other carers blind to allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Modified minimally invasive surgery alone (Experimental): Modified minimally invasive surgery alone for access and debridement of intrabony defect. This approach maximises wound stability. No application of regenerative biomaterial.
  Interventions: Procedure: Modified minimally invasive surgery
- Modified minimally invasive surgery with enamel matrix derivative (Active Comparator): Modified minimally invasive surgery access and debridement of intrabony defect combined with local application of enamel matrix derivative (regenerative biomaterial)
  Interventions: Procedure: Modified minimally invasive surgery; Procedure: Modified minimally invasive surgery with enamel matrix derivative
- Modified minimally invasive surgery with enamel matrix derivative and bone replacement graft (Active Comparator): Modified minimally invasive surgery access and debridement of intrabony defect combined with local application of enamel matrix derivative and bone replacement graft (regenerative biomaterial)
  Interventions: Procedure: Modified minimally invasive surgery; Procedure: Modified minimally invasive surgery with enamel matrix derivative; Procedure: Modified minimally invasive surgery with enamel matrix derivative and bone replacement graft

INTERVENTIONS:
Procedure: Modified minimally invasive surgery — Surgical intervention alone
  Other Names: M-MIST
Procedure: Modified minimally invasive surgery with enamel matrix derivative — Surgical intervention with local application of regenerative biomaterial
  Other Names: M-MIST with EMD
  Arms: Modified minimally invasive surgery with enamel matrix derivative; Modified minimally invasive surgery with enamel matrix derivative and bone replacement graft
Procedure: Modified minimally invasive surgery with enamel matrix derivative and bone replacement graft — Surgical intervention with local application of regenerative biomaterial and bone replacement graft
  Other Names: M-MIST EMD+BRG
  Arms: Modified minimally invasive surgery with enamel matrix derivative and bone replacement graft

SUMMARY:
Evaluate the 10-year stability clinical, radiographic outcomes obtained with the application of the modified minimally invasive surgery to deep pockets associated with intrabony defects.

DETAILED DESCRIPTION:
This 10-year follow-up of a randomized controlled clinical trial (Cortellini & Tonetti 2011) compares three treatment modalities in deep intrabony defects: i) a control group was treated with modified minimally invasive surgical technique alone (M-MIST, N=15); ii) a second group was treated with M-MIST combined with enamel matrix derivative (M-MIST EMD, N=15, Straumann, Switzerland); iii) a third group was treated with M-MIST+EMD plus Bone Mineral Derived Xenograph (M-MIST+EMD+BMDX, N=15, Geistlich, Switzerland) . The design of the original trial has been reported along with the one-year results and the details of randomization and allocation concealment (Cortellini & Tonetti 2011). Clinical outcomes of the three groups were longitudinally followed for 10 years. The 10-year follow-up was approved by the local ethical committee for clinical research of the Health Service of Tuscany (University Hospital of Firenze protocol ATRO2019, registration n° 15106_oss). All patients gave informed consent to participate into the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with periodontitis
* Presence of one intrabony defect not extending into furcation
* Good general health
* Adequate plaque control

Exclusion Criteria:

* Furcation involvement in the experimental tooth
* Inadequate control of periodontitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2009-12-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Clinical attachment level changes | 10 years
  Periodontal probing to the nearest millimetre

SECONDARY OUTCOMES:
Probing pocket depts | 10 years
  Periodontal maintainability
Tooth survival | 10 years
  Survival of treated teeth - Kaplan Mayer
Complication-free survival | 10 years
  Survival until first episode of recurrence requiring re-treatment
Cost of recurrence | 10 years
  Total cost of managing the regretted teeth including treatment of recurrence
Radiographic bone level | 10 years
  Changes in level of bone supporting the tooth

CONTACTS AND LOCATIONS:
Overall Officials: Pierpaolo Cortellini, MD, Principal Investigator — ATRO - ERGOPERIO
Locations (1):
- Studio Cortellini, Florence, Italy

IPD SHARING:
Plan to Share IPD: No
No plan to share data